CLINICAL TRIAL: NCT06700499
Title: A Multicenter, Open Label Phase II Clinical Study to Evaluate the Efficacy and Safety of AK120 in the Treatment of Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of AK120 in Subjects With Moderate to Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK120-207
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK120 300mg Q2W(Double the initial dose) (Experimental): AK120 600mg (first day) then 300mg Q2W SC until week 14.
  Interventions: Drug: AK120 300mg Q2W (JAK inhibitor users need to double the initial dose)

INTERVENTIONS:
Drug: AK120 300mg Q2W (JAK inhibitor users need to double the initial dose) — AK120 300mg Q2W SC until week 14(JAK inhibitor users need to receive a first dose of 600mg SC)

SUMMARY:
This is a multicenter, open label phase II clinical study to evaluate the efficacy and safety of AK120 in the treatment of subjects with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This is a multicenter, open label phase II clinical study to evaluate the efficacy and safety of AK120 in the treatment of subjects with moderate to severe atopic dermatitis. The total duration of the study (including screening period, treatment period and follow-up period) planned for each subject is approximately 25 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18≤75 years old.
2. Atopic dermatitis (AD) diagnosed at least half a year before screening.
3. Subject with EASI score ≥16, IGA ≥ 3, BSA ≥ 10% at screening and baseline.
4. Subjects who are suitable for continue using biological treatment assessed by investigator

Exclusion Criteria:

1. Acute onset of AD within 4 weeks before drug administration.
2. The accompany disease have been assessed by the investigators during screening period as unsuitable for participation in this study.
3. Any history or symptoms of malignant tumors in any organ within 5 years prior to screening, regardless of whether treatment has been received and whether there are signs of recurrence or metastasis
4. Have a known or suspected history of immunosuppressive diseases, including a history of invasive infections.
5. Having undergone or planned major surgery within 4 weeks prior to drug administration, or unable to fully recover from surgery prior to drug administration.
6. any medical or psychological condition that puts subjects at risk or may affect the study results assessed by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-11-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | through study completion, an average of 25 weeks
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) score | baseline to week 20
  Percentage change in EASI score from baseline. EASI score is to assesses the extent and severity of eczema in four body regions with the score ranges from 0 to 72. The higher the score, the more severe the eczema.
Investigator's Global Assessment (IGA) 0/1 | from baseline to week 20
  Percentage of subjects who achieved 0/1 in the IGA. The IGA is an assessment instrument used in clinical studies to rate the severity of atopic dermatitis globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Affected body surface area (BSA) score | from baseline to week 20
  Percentage change in BSA score from baseline. Body surface area affected by atopic dermatitis will be assessed for each section of the body (0-100%) and will be reported as a percentage of all major body sections combined.
Area under the curve(AUC) of AK120 | before drug administration at week 0/4/8/12/16
  Assessment of AUC of AK120.
Anti-drug antibodies (ADA) of AK120 | before drug administration at week 0/4/8/16/20
  Percentage of subjects with detectable anti drug antibodies (ADA) of AK120.

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Beijing Luhe Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xiyuan Hospital of CACMS, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - The Second Hospital & Clinical Medical School, Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial Dermatology Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Second people's Hospital of Shenzhen, Shenzhen, Guangdong
  - Shenzhen Hospital of University of Hong Kong, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Shijiazhuang Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People Hospital of Xingtai, Xingtai, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Anyang District Hospital, Anyang, Henan
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - Changde First People's Hospital, Changde, Hunan
  - XiangYa Hospital CentralSouth University, Changsha, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical College, Hohhot, Inner Mongolia
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Affiliated Hospital of Yanbian University Yanbian Hospital, Yanbian, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong First Medical University Affiliated Dermatology Hospital, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Shanghai Yueyang Integrated Traditional Chinese Medicine and Western Medicine Hospital, Shanghai, Shanghai Municipality
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Municipal People's Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Qujing No.1 Hospital, Qujing, Yunnan
  - Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No